CLINICAL TRIAL: NCT03964480
Title: Prospective Observational International Registry of Patients With Newly Diagnosed Peripheral T Cell Lymphoma.
Status: Recruiting | Type: Observational
Sponsor: Associazione Angela Serra per la ricerca sul cancro (Other)
Responsible Party: Sponsor
Other Study IDs: T-Cell Project 2.0
Record Dates: First submitted 2019-05-24; First posted 2019-05-28 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-02

CONDITIONS: Peripheral T-Cell Lymphoma
Keywords: Peripheral T-Cell Lymphoma; Prognosis; Outcome; Biological Characteristics; Heterogeneity; Rare Diseases
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Formalin-fixed tissue for central diagnostic pathology review; Peripheral blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study T-Cell Project 2.0 is based on the former International PTCL study designed by the International T-cell Non-Hodgkin's Lymphoma Study Group (T-Cell Project 1.0: Prospective Collection of Data in Patients With Peripheral T-Cell Lymphoma) as a prospective collection of data to predict the prognosis of patients with the more frequent subtypes of PTCL. It is a prospective, longitudinal, international, observational study of patients with newly diagnosed peripheral T-cell lymphoma aiming to verify whether this prospective collection of data would allow achieving a more accurate information on T-cell lymphomas.

The study aims to better define the clinical relevance of the new WHO Classification, the role of FDG-PET in staging and response assessment, the prognosis of different entities, the genomic landscape of different subtypes, and to investigate on most optimal treatment strategies for these neoplasms in the real-world population as well as molecular markers and to explore the prognostic or predictive implications of them in PTCL.

The study aims to better define the clinical relevance of the new WHO Classification, the role of FDG-PET in staging and response assessment, the prognosis of different entities, the genomic landscape of different subtypes, and to investigate on most optimal treatment strategies for these neoplasms in the real-world population.

DETAILED DESCRIPTION:
Peripheral T-cell non-Hodgkin lymphomas (PTCLs) are a heterogeneous group of lymphoproliferative disorder arising from mature T cells of post-thymic origin at different stages of differentiation with different morphological patterns, phenotypes, and clinical presentation. All subtypes are found more commonly in male patients, and the median age at diagnosis is 62 years. This disease is generally associated with high relapse rates and a poor prognosis, with inferior treatment outcomes compared with B-cell lymphomas and have a 5-year-survival < 32%.

T-cell lymphomas are widely recognized as a complex and heterogeneous group of lymphoproliferative disorders, generally associated with high relapse rates and a poor prognosis. Because of their rarity, they are still very poorly understood.

The introduction of new and more effective therapies and better technologies led the International T-cell non-Hodgkin's Lymphoma Study Group to launch the T-cell Project 2.0 in order to have a contemporary, real-time understanding of the T-cell lymphoma biology and treatment, together with the application of contemporary technologies to further identification of new therapeutic targets.

Per protocol, patients are evaluated according to the treating physician's standard practice. There are no specific evaluations or visits required for the Registry. Data captured in the Registry reflects what is routinely collected for patients with PTCL.

The study plans to collect the tissue sample for central review. The ordinary fixation, cryopreservation and routine tumor cytogenetics are planned for biopsy samples. Chairmen of the Histopathology Review Panel will locate Regional sites where expert hematopathologists will review the material and perform a panel of immunostains (T-cell panel + CD20) and markers not assessed at local site.

Adding of blood sample collection will allow estimating prospectively the frequency of pEBVd detection in our cohort of PTCL patients at baseline and at the end of initial therapy, to characterize agreement between pEBVd and EBER in tumor tissue, and to explore the prognostic or predictive implications of detectable pEBVd in PTCL. Finally, to investigate the genetics and pathogenic mechanisms of aggressive PTCLs on an international scale.

ELIGIBILITY:
Inclusion Criteria:

1. Previously-untreated patients with de novo diagnosis of peripheral T-cell or NK/T-cell lymphoma:

   * T-cell large granular lymphocytic leukaemia;
   * Chronic lymphoproliferative disorder of NK cells;
   * Aggressive NK-cell leukaemia;
   * Adult T-cell leukaemia/lymphoma;
   * Extranodal NK/T-cell lymphoma, nasal type;
   * Intestinal T-cell lymphoma;
   * Hepatosplenic T-cell lymphoma;
   * Subcutaneous panniculitis-like T-cell lymphoma;
   * Peripheral T-cell lymphoma, not otherwise specified;
   * Angioimmunoblastic T-cell lymphoma and other nodal lymphomas of T follicular helper cell origin;
   * Anaplastic large cell lymphoma, ALK-positive;
   * Anaplastic large cell lymphoma, ALK-negative;
   * Breast implant-associated anaplastic large cell lymphoma.
2. Age 18 and over;
3. Tissue biopsy adequate for diagnosis and classification and available for centralized review;
4. Clinical data including baseline information on disease localization and laboratory parameters at staging, features of treatment adopted and assurance of follow-up updating for at least 2 years are requested;
5. Written informed consent.

Exclusion Criteria:

1. Diagnosis of:

   * EBV-positive T-cell and NK-cell lymphoproliferative diseases of childhood
   * Mycosis fungoides;
   * Sézary syndrome;
   * Primary cutaneous CD30-positive T-cell lymphoproliferative disorders;
   * Primary cutaneous peripheral T-cell lymphomas, rare subtypes;
   * T-cell lymphoblastic lymphoma/leukemia
   * T-cell prolymphocitic leukemia
2. Age < 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously-untreated patients with de novo diagnosis of peripheral T-cell or NK/T-cell lymphoma:
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-10-14 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2 year
  Measured from the date of diagnosis until the date of disease progression or death from T-cell Lymphoma

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 and 5 year
  Measured from the date of diagnosis until death from any cause
Progression-Free Survival (PFS) | 3 and 5 years
  Measured from the date of diagnosis until the date of disease progression or death from T-cell Lymphoma
Event Free Survival (EFS) | at 24 months
  Measured from the date of diagnosis until the date of event
Complete Response Rate (CR) | at 30 months
  Complete response rate at 30 months (CR30) after enrollment (i.e., initiation of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Federico, MD, Study Director — University of Modena and Reggio Emilia, Centro Oncologico Modenese, Modena, Italy; Attilio Guarini, MD, Principal Investigator — U.O. Ematologia, IRCCS Istituto Tumori "Giovanni Paolo II"; Julie Vose, MD, Principal Investigator — Section of Hematology/Oncology, Nebraska Medical Center, USA; Steven Horwitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Miles Prince, MD, Principal Investigator — Peter MacCallum Cancer Center, Melbourne, Australia; Kim Won Seog, MD, Principal Investigator — Hematology-Oncology Samsung Medical Center, Seoul, South Korea; Dolores Caballero, MD, Principal Investigator — Instituto Biosanitaria de Salamanca, Salamanca, Spain; Francesco Zaya, MD, Principal Investigator — Azienda Sanitaria Universitaria Integrata S.M. Misericordia, Udine, Italy; Stefano Luminari, MD, Principal Investigator — S.C. Ematologia, Arcispedale S. Maria Nuova-IRCCS, Reggio Emilia, Italy; Ranjana Advani, MD, Principal Investigator — Stanford University Medical Center, Stanford, CA, USA; Andrei Shustov, MD, Principal Investigator — Seattle Cancer Care Alliance, Seattle, WA, USA; Pierluigi Porcu, MD, Principal Investigator — Hematopoietic Stem Cell Transplantation, Sidney Kimmel Cancer Center, USA; Astrid Pavlovsky, MD, Principal Investigator — Centro de Hematologia, FUNDALEU, Buenos Aires, Argentina; Carlos Chiattone, MD, Principal Investigator — Departamento de Clinica Médica, FCM da Santa Casa de Sao Paulo, Sao Paulo, Brazil; Francine Foss, MD, Principal Investigator — Yale University School of Medicine, New Haven, CT, USA; Christopher Fox, MD, Principal Investigator — Clinical Haematology, Nottingham University Hospitals NHS Trust, Nottingham, UK
Locations (6):
- Stanford University, Stanford, California, United States
- Italy (3):
  - IRCCS Istituto Tumori "Giovanni Paolo II", Bari
  - Palermo_La Maddalena, Palermo
  - Terni-Santa Maria, Terni
- Cluj Napoca_Ion Chiricuta Oncology Institute, Cluj-Napoca, Romania
- National Cancer Institute, Kiev, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
We plan to share with other involved researchers the minimum information on IPD for publication.
Time Frame: Preliminary analysis results will be made available during the study on the single population and separately for each sub-type. Final results will be made available 6-12 months after the end of the study.

REFERENCES:
- [Background] Ansell S. How to select the frontline treatment for a patient with peripheral T-cell lymphoma. Leuk Lymphoma. 2016;57(4):783-8. doi: 10.3109/10428194.2016.1140760. Epub 2016 Feb 5. PMID 26850659
- [Background] Vose J, Armitage J, Weisenburger D; International T-Cell Lymphoma Project. International peripheral T-cell and natural killer/T-cell lymphoma study: pathology findings and clinical outcomes. J Clin Oncol. 2008 Sep 1;26(25):4124-30. doi: 10.1200/JCO.2008.16.4558. Epub 2008 Jul 14. PMID 18626005
- [Background] A clinical evaluation of the International Lymphoma Study Group classification of non-Hodgkin's lymphoma. The Non-Hodgkin's Lymphoma Classification Project. Blood. 1997 Jun 1;89(11):3909-18. PMID 9166827
- [Background] Savage KJ. Peripheral T-cell lymphomas. Blood Rev. 2007 Jul;21(4):201-16. doi: 10.1016/j.blre.2007.03.001. Epub 2007 May 18. PMID 17512649
- [Background] Iqbal J, Wright G, Wang C, Rosenwald A, Gascoyne RD, Weisenburger DD, Greiner TC, Smith L, Guo S, Wilcox RA, Teh BT, Lim ST, Tan SY, Rimsza LM, Jaffe ES, Campo E, Martinez A, Delabie J, Braziel RM, Cook JR, Tubbs RR, Ott G, Geissinger E, Gaulard P, Piccaluga PP, Pileri SA, Au WY, Nakamura S, Seto M, Berger F, de Leval L, Connors JM, Armitage J, Vose J, Chan WC, Staudt LM; Lymphoma Leukemia Molecular Profiling Project and the International Peripheral T-cell Lymphoma Project. Gene expression signatures delineate biological and prognostic subgroups in peripheral T-cell lymphoma. Blood. 2014 May 8;123(19):2915-23. doi: 10.1182/blood-2013-11-536359. Epub 2014 Mar 14. PMID 24632715
- [Background] Barbui T, Thiele J, Gisslinger H, Kvasnicka HM, Vannucchi AM, Guglielmelli P, Orazi A, Tefferi A. The 2016 WHO classification and diagnostic criteria for myeloproliferative neoplasms: document summary and in-depth discussion. Blood Cancer J. 2018 Feb 9;8(2):15. doi: 10.1038/s41408-018-0054-y. PMID 29426921
- [Background] Foss FM, Zinzani PL, Vose JM, Gascoyne RD, Rosen ST, Tobinai K. Peripheral T-cell lymphoma. Blood. 2011 Jun 23;117(25):6756-67. doi: 10.1182/blood-2010-05-231548. Epub 2011 Apr 14. PMID 21493798
- [Background] Weisenburger DD, Savage KJ, Harris NL, Gascoyne RD, Jaffe ES, MacLennan KA, Rudiger T, Pileri S, Nakamura S, Nathwani B, Campo E, Berger F, Coiffier B, Kim WS, Holte H, Federico M, Au WY, Tobinai K, Armitage JO, Vose JM; International Peripheral T-cell Lymphoma Project. Peripheral T-cell lymphoma, not otherwise specified: a report of 340 cases from the International Peripheral T-cell Lymphoma Project. Blood. 2011 Mar 24;117(12):3402-8. doi: 10.1182/blood-2010-09-310342. Epub 2011 Jan 26. PMID 21270441
- [Background] Gallamini A, Stelitano C, Calvi R, Bellei M, Mattei D, Vitolo U, Morabito F, Martelli M, Brusamolino E, Iannitto E, Zaja F, Cortelazzo S, Rigacci L, Devizzi L, Todeschini G, Santini G, Brugiatelli M, Federico M; Intergruppo Italiano Linfomi. Peripheral T-cell lymphoma unspecified (PTCL-U): a new prognostic model from a retrospective multicentric clinical study. Blood. 2004 Apr 1;103(7):2474-9. doi: 10.1182/blood-2003-09-3080. Epub 2003 Nov 26. PMID 14645001
- [Background] Went P, Agostinelli C, Gallamini A, Piccaluga PP, Ascani S, Sabattini E, Bacci F, Falini B, Motta T, Paulli M, Artusi T, Piccioli M, Zinzani PL, Pileri SA. Marker expression in peripheral T-cell lymphoma: a proposed clinical-pathologic prognostic score. J Clin Oncol. 2006 Jun 1;24(16):2472-9. doi: 10.1200/JCO.2005.03.6327. Epub 2006 Apr 24. PMID 16636342
- [Background] Lage LA, Cabral TC, Costa Rde O, Goncalves Mde C, Levy D, Zerbini MC, Pereira J. Primary nodal peripheral T-cell lymphomas: diagnosis and therapeutic considerations. Rev Bras Hematol Hemoter. 2015 Jul-Aug;37(4):277-84. doi: 10.1016/j.bjhh.2015.03.017. Epub 2015 Jun 7. PMID 26190436
- [Background] Dearden CE, Johnson R, Pettengell R, Devereux S, Cwynarski K, Whittaker S, McMillan A; British Committee for Standards in Haematology. Guidelines for the management of mature T-cell and NK-cell neoplasms (excluding cutaneous T-cell lymphoma). Br J Haematol. 2011 May;153(4):451-85. doi: 10.1111/j.1365-2141.2011.08651.x. Epub 2011 Apr 11. PMID 21480860
- [Background] Karakas T, Bergmann L, Stutte HJ, Jager E, Knuth A, Weidmann E, Mitrou PS, Hoelzer D. Peripheral T-cell lymphomas respond well to vincristine, adriamycin, cyclophosphamide, prednisone and etoposide (VACPE) and have a similar outcome as high-grade B-cell lymphomas. Leuk Lymphoma. 1996 Dec;24(1-2):121-9. doi: 10.3109/10428199609045720. PMID 9049968
- [Background] Schmitz N, Trumper L, Ziepert M, Nickelsen M, Ho AD, Metzner B, Peter N, Loeffler M, Rosenwald A, Pfreundschuh M. Treatment and prognosis of mature T-cell and NK-cell lymphoma: an analysis of patients with T-cell lymphoma treated in studies of the German High-Grade Non-Hodgkin Lymphoma Study Group. Blood. 2010 Nov 4;116(18):3418-25. doi: 10.1182/blood-2010-02-270785. Epub 2010 Jul 21. PMID 20660290
- [Background] d'Amore F, Gaulard P, Trumper L, Corradini P, Kim WS, Specht L, Bjerregaard Pedersen M, Ladetto M; ESMO Guidelines Committee. Peripheral T-cell lymphomas: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2015 Sep;26 Suppl 5:v108-15. doi: 10.1093/annonc/mdv201. No abstract available. PMID 26314772
- [Background] Dreyling M, Thieblemont C, Gallamini A, Arcaini L, Campo E, Hermine O, Kluin-Nelemans JC, Ladetto M, Le Gouill S, Iannitto E, Pileri S, Rodriguez J, Schmitz N, Wotherspoon A, Zinzani P, Zucca E. ESMO Consensus conferences: guidelines on malignant lymphoma. part 2: marginal zone lymphoma, mantle cell lymphoma, peripheral T-cell lymphoma. Ann Oncol. 2013 Apr;24(4):857-77. doi: 10.1093/annonc/mds643. Epub 2013 Feb 20. PMID 23425945
- [Background] Reddy NM, Evens AM. Chemotherapeutic advancements in peripheral T-cell lymphoma. Semin Hematol. 2014 Jan;51(1):17-24. doi: 10.1053/j.seminhematol.2013.11.006. Epub 2013 Nov 14. PMID 24468312
- [Background] Cheah CY, Oki Y, Fanale MA. Novel treatments for T-cell lymphoma. Am Soc Clin Oncol Educ Book. 2015:e468-78. doi: 10.14694/EdBook_AM.2015.35.e468. PMID 25993211
- [Background] Enblad G, Hagberg H, Erlanson M, Lundin J, MacDonald AP, Repp R, Schetelig J, Seipelt G, Osterborg A. A pilot study of alemtuzumab (anti-CD52 monoclonal antibody) therapy for patients with relapsed or chemotherapy-refractory peripheral T-cell lymphomas. Blood. 2004 Apr 15;103(8):2920-4. doi: 10.1182/blood-2003-10-3389. Epub 2003 Dec 30. PMID 15070664
- [Background] Zinzani PL, Alinari L, Tani M, Fina M, Pileri S, Baccarani M. Preliminary observations of a phase II study of reduced-dose alemtuzumab treatment in patients with pretreated T-cell lymphoma. Haematologica. 2005 May;90(5):702-3. PMID 15921394
- [Background] Zinzani PL, Venturini F, Stefoni V, Fina M, Pellegrini C, Derenzini E, Gandolfi L, Broccoli A, Argnani L, Quirini F, Pileri S, Baccarani M. Gemcitabine as single agent in pretreated T-cell lymphoma patients: evaluation of the long-term outcome. Ann Oncol. 2010 Apr;21(4):860-863. doi: 10.1093/annonc/mdp508. Epub 2009 Nov 3. PMID 19887465
- [Background] Zinzani PL, Musuraca G, Tani M, Stefoni V, Marchi E, Fina M, Pellegrini C, Alinari L, Derenzini E, de Vivo A, Sabattini E, Pileri S, Baccarani M. Phase II trial of proteasome inhibitor bortezomib in patients with relapsed or refractory cutaneous T-cell lymphoma. J Clin Oncol. 2007 Sep 20;25(27):4293-7. doi: 10.1200/JCO.2007.11.4207. Epub 2007 Aug 20. PMID 17709797
- [Background] Toumishey E, Prasad A, Dueck G, Chua N, Finch D, Johnston J, van der Jagt R, Stewart D, White D, Belch A, Reiman T. Final report of a phase 2 clinical trial of lenalidomide monotherapy for patients with T-cell lymphoma. Cancer. 2015 Mar 1;121(5):716-23. doi: 10.1002/cncr.29103. Epub 2014 Oct 29. PMID 25355245
- [Background] Morschhauser F, Fitoussi O, Haioun C, Thieblemont C, Quach H, Delarue R, Glaisner S, Gabarre J, Bosly A, Lister J, Li J, Coiffier B. A phase 2, multicentre, single-arm, open-label study to evaluate the safety and efficacy of single-agent lenalidomide (Revlimid) in subjects with relapsed or refractory peripheral T-cell non-Hodgkin lymphoma: the EXPECT trial. Eur J Cancer. 2013 Sep;49(13):2869-76. doi: 10.1016/j.ejca.2013.04.029. Epub 2013 May 31. PMID 23731832
- [Background] O'Connor OA, Horwitz S, Hamlin P, Portlock C, Moskowitz CH, Sarasohn D, Neylon E, Mastrella J, Hamelers R, Macgregor-Cortelli B, Patterson M, Seshan VE, Sirotnak F, Fleisher M, Mould DR, Saunders M, Zelenetz AD. Phase II-I-II study of two different doses and schedules of pralatrexate, a high-affinity substrate for the reduced folate carrier, in patients with relapsed or refractory lymphoma reveals marked activity in T-cell malignancies. J Clin Oncol. 2009 Sep 10;27(26):4357-64. doi: 10.1200/JCO.2008.20.8470. Epub 2009 Aug 3. PMID 19652067
- [Background] O'Connor OA, Pro B, Pinter-Brown L, Bartlett N, Popplewell L, Coiffier B, Lechowicz MJ, Savage KJ, Shustov AR, Gisselbrecht C, Jacobsen E, Zinzani PL, Furman R, Goy A, Haioun C, Crump M, Zain JM, Hsi E, Boyd A, Horwitz S. Pralatrexate in patients with relapsed or refractory peripheral T-cell lymphoma: results from the pivotal PROPEL study. J Clin Oncol. 2011 Mar 20;29(9):1182-9. doi: 10.1200/JCO.2010.29.9024. Epub 2011 Jan 18. PMID 21245435
- [Background] Damaj G, Gressin R, Bouabdallah K, Cartron G, Choufi B, Gyan E, Banos A, Jaccard A, Park S, Tournilhac O, Schiano-de Collela JM, Voillat L, Joly B, Le Gouill S, Saad A, Cony-Makhoul P, Vilque JP, Sanhes L, Schmidt-Tanguy A, Bubenheim M, Houot R, Diouf M, Marolleau JP, Bene MC, Martin A, Lamy T. Results from a prospective, open-label, phase II trial of bendamustine in refractory or relapsed T-cell lymphomas: the BENTLY trial. J Clin Oncol. 2013 Jan 1;31(1):104-10. doi: 10.1200/JCO.2012.43.7285. Epub 2012 Oct 29. PMID 23109692
- [Background] Piekarz RL, Frye R, Prince HM, Kirschbaum MH, Zain J, Allen SL, Jaffe ES, Ling A, Turner M, Peer CJ, Figg WD, Steinberg SM, Smith S, Joske D, Lewis I, Hutchins L, Craig M, Fojo AT, Wright JJ, Bates SE. Phase 2 trial of romidepsin in patients with peripheral T-cell lymphoma. Blood. 2011 Jun 2;117(22):5827-34. doi: 10.1182/blood-2010-10-312603. Epub 2011 Feb 25. PMID 21355097
- [Background] Suwiwat S, Pradutkanchana J, Ishida T, Mitarnun W. Quantitative analysis of cell-free Epstein-Barr virus DNA in the plasma of patients with peripheral T-cell and NK-cell lymphomas and peripheral T-cell proliferative diseases. J Clin Virol. 2007 Dec;40(4):277-83. doi: 10.1016/j.jcv.2007.08.013. Epub 2007 Nov 9. PMID 17996493
- [Background] Kim YR, Kim SJ, Cheong JW, Chung H, Jang JE, Kim Y, Yang WI, Min YH, Kim JS. Pretreatment Epstein-Barr virus DNA in whole blood is a prognostic marker in peripheral T-cell lymphoma. Oncotarget. 2017 Sep 23;8(54):92312-92323. doi: 10.18632/oncotarget.21251. eCollection 2017 Nov 3. PMID 29190917
- [Background] Lynch RC, Gratzinger D, Advani RH. Clinical Impact of the 2016 Update to the WHO Lymphoma Classification. Curr Treat Options Oncol. 2017 Jul;18(7):45. doi: 10.1007/s11864-017-0483-z. PMID 28670664
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Background] Vittinghoff E, McCulloch CE. Relaxing the rule of ten events per variable in logistic and Cox regression. Am J Epidemiol. 2007 Mar 15;165(6):710-8. doi: 10.1093/aje/kwk052. Epub 2006 Dec 20. PMID 17182981
- [Background] Ogundimu EO, Altman DG, Collins GS. Adequate sample size for developing prediction models is not simply related to events per variable. J Clin Epidemiol. 2016 Aug;76:175-82. doi: 10.1016/j.jclinepi.2016.02.031. Epub 2016 Mar 8. PMID 26964707
- [Background] Harrell FE Jr, Lee KL, Mark DB. Multivariable prognostic models: issues in developing models, evaluating assumptions and adequacy, and measuring and reducing errors. Stat Med. 1996 Feb 28;15(4):361-87. doi: 10.1002/(SICI)1097-0258(19960229)15:43.0.CO;2-4. PMID 8668867
- [Background] Royston P, Sauerbrei W. A new measure of prognostic separation in survival data. Stat Med. 2004 Mar 15;23(5):723-48. doi: 10.1002/sim.1621. PMID 14981672
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Coiffier B, Pro B, Prince HM, Foss F, Sokol L, Greenwood M, Caballero D, Borchmann P, Morschhauser F, Wilhelm M, Pinter-Brown L, Padmanabhan S, Shustov A, Nichols J, Carroll S, Balser J, Balser B, Horwitz S. Results from a pivotal, open-label, phase II study of romidepsin in relapsed or refractory peripheral T-cell lymphoma after prior systemic therapy. J Clin Oncol. 2012 Feb 20;30(6):631-6. doi: 10.1200/JCO.2011.37.4223. Epub 2012 Jan 23. PMID 22271479
- [Background] Coiffier B, Pro B, Prince HM, Foss F, Sokol L, Greenwood M, Caballero D, Morschhauser F, Wilhelm M, Pinter-Brown L, Padmanabhan Iyer S, Shustov A, Nielsen T, Nichols J, Wolfson J, Balser B, Horwitz S. Romidepsin for the treatment of relapsed/refractory peripheral T-cell lymphoma: pivotal study update demonstrates durable responses. J Hematol Oncol. 2014 Jan 23;7:11. doi: 10.1186/1756-8722-7-11. PMID 24456586
- [Background] Pro B, Advani R, Brice P, Bartlett NL, Rosenblatt JD, Illidge T, Matous J, Ramchandren R, Fanale M, Connors JM, Yang Y, Sievers EL, Kennedy DA, Shustov A. Brentuximab vedotin (SGN-35) in patients with relapsed or refractory systemic anaplastic large-cell lymphoma: results of a phase II study. J Clin Oncol. 2012 Jun 20;30(18):2190-6. doi: 10.1200/JCO.2011.38.0402. Epub 2012 May 21. PMID 22614995
- [Background] Horwitz SM, Advani RH, Bartlett NL, Jacobsen ED, Sharman JP, O'Connor OA, Siddiqi T, Kennedy DA, Oki Y. Objective responses in relapsed T-cell lymphomas with single-agent brentuximab vedotin. Blood. 2014 May 15;123(20):3095-100. doi: 10.1182/blood-2013-12-542142. Epub 2014 Mar 20. PMID 24652992
- [Background] Foss F, Advani R, Duvic M, Hymes KB, Intragumtornchai T, Lekhakula A, Shpilberg O, Lerner A, Belt RJ, Jacobsen ED, Laurent G, Ben-Yehuda D, Beylot-Barry M, Hillen U, Knoblauch P, Bhat G, Chawla S, Allen LF, Pohlman B. A Phase II trial of Belinostat (PXD101) in patients with relapsed or refractory peripheral or cutaneous T-cell lymphoma. Br J Haematol. 2015 Mar;168(6):811-9. doi: 10.1111/bjh.13222. Epub 2014 Nov 17. PMID 25404094
- [Background] O'Connor OA, Horwitz S, Masszi T, Van Hoof A, Brown P, Doorduijn J, Hess G, Jurczak W, Knoblauch P, Chawla S, Bhat G, Choi MR, Walewski J, Savage K, Foss F, Allen LF, Shustov A. Belinostat in Patients With Relapsed or Refractory Peripheral T-Cell Lymphoma: Results of the Pivotal Phase II BELIEF (CLN-19) Study. J Clin Oncol. 2015 Aug 10;33(23):2492-9. doi: 10.1200/JCO.2014.59.2782. Epub 2015 Jun 22. PMID 26101246
- [Background] Bellei M, Sabattini E, Pesce EA, Ko YH, Kim WS, Cabrera ME, Martinez V, Dlouhy I, Paes RP, Barrese T, Vassallo J, Tarantino V, Vose J, Weisenburger D, Rudiger T, Federico M, Pileri S. Pitfalls and major issues in the histologic diagnosis of peripheral T-cell lymphomas: results of the central review of 573 cases from the T-Cell Project, an international, cooperative study. Hematol Oncol. 2017 Dec;35(4):630-636. doi: 10.1002/hon.2316. Epub 2016 Jun 3. PMID 27255982
- [Background] Boddicker RL, Razidlo GL, Feldman AL. Genetic alterations affecting GTPases and T-cell receptor signaling in peripheral T-cell lymphomas. Small GTPases. 2019 Jan;10(1):33-39. doi: 10.1080/21541248.2016.1263718. Epub 2017 Jan 6. PMID 27898263
- [Background] Haverkos BM, Huang Y, Gru A, Pancholi P, Freud AG, Mishra A, Ruppert AS, Baiocchi RA, Porcu P. Frequency and clinical correlates of elevated plasma Epstein-Barr virus DNA at diagnosis in peripheral T-cell lymphomas. Int J Cancer. 2017 Apr 15;140(8):1899-1906. doi: 10.1002/ijc.30566. PMID 27943278